CLINICAL TRIAL: NCT01125410
Title: Phase III Comparative Study of Efficacy of 10 mg Dequalinium Chloride (Fluomizin) in the Local Treatment of Bacterial Vaginosis
Brief Title: Comparative Study of Efficacy of 10 mg Dequalinium Chloride (Fluomizin) in the Local Treatment of Bacterial Vaginosis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Medinova AG (Industry)
Responsible Party: Dr. Philipp Grob, Medinova AG
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Med380104
Record Dates: First submitted 2010-05-11; First posted 2010-05-18 (Estimated); Last update posted 2010-05-18 (Estimated); Status verified 2010-05

CONDITIONS: Bacterial Vaginosis
Keywords: Fluomizin; Dequalinium chloride; Bacterial vaginosis; vaginal therapy
MeSH Terms: conditions — Vaginosis, Bacterial | interventions — Dequalinium; Clindamycin

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Dequalinium chloride 10mg (Experimental)
  Interventions: Drug: Dequalinium chloride
- clindamycin vaginal cream 2% (Active Comparator)
  Interventions: Drug: Clindamycin

INTERVENTIONS:
Drug: Dequalinium chloride — Vaginal tablet, 10mg, 1 tablet daily for 6 days
  Arms: Dequalinium chloride 10mg
Drug: Clindamycin — vaginal cream, 2%, once daily for 7 days
  Arms: clindamycin vaginal cream 2%

SUMMARY:
The purpose of this clinical study was to evaluate whether vaginal tablets containing 10 mg dequalinium chloride (Fluomizin) are comparable in clinical efficacy and safety to clindamycin vaginal cream (2%) in patients suffering from bacterial vaginosis.

DETAILED DESCRIPTION:
An international, multi-center, single-blind, randomized, active-controlled study with two parallel groups in patients with bacterial vaginosis. Eligible patients were randomized to receive Fluomizin vaginal tablets for 6 days or Clindamycin vaginal cream (2%) for 7 days. Control examinations were performed 3 to 14 days and 2 to 6 weeks after the end of the therapy.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of bacterial vaginosis
* Women aged 18-55 years

Exclusion Criteria:

* Pregnancy or lactation
* Uterine bleeding (including menstruation but not including cervical contact bleeding on sampling) or vaginal bleeding of unknown origin
* Acute infections of the upper genital tract
* Clinical Symptoms of a vulvovaginal Candidiasis
* Use of anti-infectives (local or systemic) in the previous 14 days and/or during the study

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 321 (Actual)
Dates: Start 2007-01; Primary Completion 2008-07 (Actual); Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
clinical cure rate | 1 week (on average)
  Clinical cure rate based on Amsel criteria. For cure, clue cells have to be negative and not more than one of the other criteria positive
Clinical cure rate | 4 weeks (on average)
  Clinical cure rate based on Amsel criteria, where cure was defined as clue cells being negative and not more than one of the other criteria positive

SECONDARY OUTCOMES:
Treatment failure | 4 weeks
  Treatment failures include non-responders and recurrences
Incidence of ADRs | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Ernst Rainer Weissenbacher, MD, Principal Investigator — Klinik und Poliklinik für Frauenheilkunde und Geburtshilfe, LMU Munich
Locations (14):
- Belgium (4):
  - AZ Imelda Ziekenhuis, Bonheiden
  - AZ St. Dimpna, Geel
  - AZ Ziekenhuis Oost-Limburg, Genk
  - AZ Heilig Hart, Tienen
- Czechia (6):
  - Centrum Ambulantni gynekologie a prodnictvi, Brno
  - Faculty Hospital Brno, Brno
  - University Hospital Hradec Kralove, Hradec Králové
  - Charles University, Prague
  - Fakultni nemocnice Na Bulovce, Prague
  - Ambulance pro gynekologie a prodnictvi, Telč
- LMU Munich, Munich, Germany
- JLF UK a MFN, Martin, Slovakia
- Switzerland (2):
  - University Hospital of Geneva and Faculty of Medicine, Geneva
  - CHUV, Lausanne

REFERENCES:
- [Derived] Weissenbacher ER, Donders G, Unzeitig V, Martinez de Tejada B, Gerber S, Halaska M, Spacek J; Fluomizin Study Group. A comparison of dequalinium chloride vaginal tablets (Fluomizin(R)) and clindamycin vaginal cream in the treatment of bacterial vaginosis: a single-blind, randomized clinical trial of efficacy and safety. Gynecol Obstet Invest. 2012;73(1):8-15. doi: 10.1159/000332398. Epub 2011 Dec 24. PMID 22205034